CLINICAL TRIAL: NCT05534776
Title: Validation of 5-Point Investigator Global Assessments for Pemphigus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Premier Specialists, Australia (Other)
Responsible Party: Principal Investigator, Dedee Murrell, Professor, Director of Premier Specialists, Premier Specialists, Australia
Other Study IDs: IGA Pemphigus
Record Dates: First submitted 2022-08-29; First posted 2022-09-09 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pemphigus
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Scoring Session: Participants whose de-identified photos will be printed in the first booklet for the first scoring session.
  Interventions: Other: Investigator Global Assessments (IGAs)
- Second Scoring Session: Participants whose de-identified photos will be printed in the second booklet for the second scoring session.
  Interventions: Other: Investigator Global Assessments (IGAs)

INTERVENTIONS:
Other: Investigator Global Assessments (IGAs) — 5-Point scale from 0-4 to score the severity of pemphigus, where 0=clear, 1=almost clear, 2=mild, 3=moderate and 4=severe.

SUMMARY:
This study aims to explore the reliability and validity of newly developed Investigator Global Assessments (IGAs) in scoring the severity of pemphigus. IGAs are simple 5-point scales ranging from clear - severe and are preferred by the FDA as endpoints in clinical trials.

DETAILED DESCRIPTION:
This study aims to obtain statistical data regarding the inter-rater and intra-rater reliability of the IGAs, Pemphigus Disease Activity Index (PDAI) and Autoimmune Bullous Skin Disease Intensity Score (ABSIS) as well as the convergent validity of the IGAs with the PDAI and objective component of the ABSIS.

Photograph sets of pemphigus lesions will be gathered from the lead site and participant sites. They will be de-identified and printed in a two hardcopy booklets; the first containing 20 photo sets and the second containing 17 new photo sets and 3 repeat photo sets. In the first part of the study, 8 dermatologists will score 20 sets of photographs of pemphigus lesions (a mixture of skin and mucosal lesions), using the IGAs for pemphigus as well as the PDAI and ABSIS. The first booklet will be mailed to dermatologists and they will use the booklet to score each photo set and will submit their scores in a confidential online survey. In the second part of the study, the second booklet will be sent to dermatologists in the same manner 4 weeks later, and each dermatologist will score the photo sets using the same scoring tools. It is estimated that each scoring session will take two hours to complete. Data gathered here will allow for calculation of inter-rater reliability and intra-rater reliability of the IGAs and convergent validity of the IGAs with PDAI and ABSIS.

Later, a sub-study will occur to calculate minimal clinically important differences (MCID) for the IGAs and PDAI. This will involve scoring pemphigus severity of patients at Premier Specialists using PDAI and IGA scores and a Likert score to classify patients as improved, stable or deteriorated compared to previous visits.

ELIGIBILITY:
Inclusion Criteria:

* Having pemphigus diagnosed by a qualified dermatologist
* Aged 18 or older at the time of photography

Exclusion Criteria:

* Those whose photographs are unable to be adequately de-identified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the special bullous clinic at the lead site's dermatology practice who have been diagnosed with pemphigus.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-21 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
IGA-PV-M (D/P/F), IGA-PV-S (D/P/F), IGA-PF (D/P/F) | Baseline
  IGA score of pemphigus severity, possible score from 0-4
Pemphigus Disease Activity Index (PDAI) Score | Baseline
  Possible score from 0-263
Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) | Baseline
  Possible score from 0-206

CONTACTS AND LOCATIONS:
Locations (7):
- Premier Specialists, Kogarah, New South Wales, Australia
- Medical University of Sofia, Sofia, Bulgaria
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Razi Hospital, Tehran, Iran
- Tel Aviv Medical Centre, Tel Aviv, Israel
- National University Hospital of Singapore, Singapore, Singapore
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided